CLINICAL TRIAL: NCT05739318
Title: The Accuracy of the Diameter of Double-lumen Tube Measured by Different Methods as a Guide to the Size Selection of Double-lumen Tube
Brief Title: the Diameter of Double-lumen Tube Measured by Different Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2022A123
Record Dates: First submitted 2023-02-09; First posted 2023-02-22 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2023-02

CONDITIONS: Therapeutic Procedural Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The cuff of endotracheal and endobronchial is collapsed (Experimental): The diameter of double-lumen tube at the cuff of endotracheal and endobronchial during the cuff is collapsed
  Interventions: Device: The cuff of endotracheal and endobronchial is collapsed
- The cuff of endotracheal and endobronchial is inflated (Experimental): The diameter of double-lumen tube at the cuff of endotracheal and endobronchial during the cuff is inflated
  Interventions: Device: The cuff of endotracheal and endobronchial is inflated

INTERVENTIONS:
Device: The cuff of endotracheal and endobronchial is collapsed — The diameter of double-lumen tube at the cuff of endotracheal and endobronchial when the cuff is collapsed as the diameter of double-lumen tube and select a double-lumen tube that matches the patient's trachea and bronchial innerdiameter based on this diameter
  Arms: The cuff of endotracheal and endobronchial is collapsed
Device: The cuff of endotracheal and endobronchial is inflated — The diameter of double-lumen tube at the cuff of endotracheal and endobronchial when the cuff is inflated as the diameter of double-lumen tube and select a double-lumen tube that matches the patient's trachea and bronchial innerdiameter based on this diameter
  Arms: The cuff of endotracheal and endobronchial is inflated

SUMMARY:
The comparison of the diameter of double-lumen tube at the cuff of endotracheal and endobronchial during the cuff was collapse or inflated as a guide for the selection of the size of double-lumen tube.

DETAILED DESCRIPTION:
The comparison of the diameter of double-lumen tube at the cuff of endotracheal and endobronchial during the cuff was collapse or inflated as a guide for the selection of the size of double-lumen tube.

ELIGIBILITY:
Inclusion Criteria:

BMI less than 35 kg/m2 ASA classifications of I-III, Modified Mallampati classification 1 or 2 Under general anesthesia

Exclusion Criteria:

Age younger than 18 yr or older than 70 yr

* ASA class IV or V
* Abnormalities of the heart, brain, liver, lung, kidney and coagulation function

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Incidence of complications | 12 weeks
  Incidence of postoperative hoarseness and throat pain in patients

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Qinhuangdao, Qinhuangdao, Hebei, China

REFERENCES:
- [Derived] Cui G, Zhao L, Chi C, Liang S, Liu Z. The feasibility and accuracy of the method for selecting the optimal size of double-lumen tube in thoracic surgery: a prospective, randomized controlled trial. Sci Rep. 2024 Jul 30;14(1):17539. doi: 10.1038/s41598-024-68349-z. PMID 39080380